CLINICAL TRIAL: NCT02178735
Title: Clinical Outcomes and Urodynamic Effects After Vaginal Tailored Mesh Surgery for Pelvic Organ Prolapse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201404024RINC
Record Dates: First submitted 2014-06-09; First posted 2014-07-01 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse, vaginal mesh, urodynamic studies
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anterior compartment prolapse (Experimental): Woman with cystocele who underwent anterior vaginal tailored mesh surgery
  Interventions: Procedure: Anterior vaginal tailored mesh surgery
- Posterior compartment prolapse (Experimental): Woman with rectocele, enterocele, uterine prolapse, vaginal stump prolpase who underwent posterior vaginal tailored mesh surgery
  Interventions: Procedure: Posterior vaginal tailored mesh surgery
- anterior and posterior prolapse (Experimental): Woman with cystocele and rectocele/uterine prolapse/vaginal vault prolapse/enterocele who underwent anterior and posterior vaginal tailored mesh surgery
  Interventions: Procedure: Anterior vaginal tailored mesh surgery; Procedure: Posterior vaginal tailored mesh surgery

INTERVENTIONS:
Procedure: Anterior vaginal tailored mesh surgery — Anterior vaginal tailored mesh surgery for repair of cystocele with or without stress urinary incontinence
  Arms: Anterior compartment prolapse; anterior and posterior prolapse
Procedure: Posterior vaginal tailored mesh surgery — Posterior vaginal tailored mesh surgery for repair of enterocele, rectocele, vaginal vault prolapse or uterine prolapse
  Arms: Posterior compartment prolapse; anterior and posterior prolapse

SUMMARY:
To evaluate the clinical outcome and urodynamic effect of two novel vaginal tailored mesh surgeries.

DETAILED DESCRIPTION:
We will review the medical records (including medical data, urodynamic data, pad weight data, etc) of women who underwent either anterior or posterior novel vaginal tailored mesh surgeries at National Taiwan University Hospital between November 2011 and November 2013.

ELIGIBILITY:
Inclusion Criteria:

* All women with pelvic organ prolapse who underwent either anterior or/and posterior vaginal tailored mesh surgeries in National Taiwan University Hospital between November 2011 and November 2013

Exclusion Criteria: nil

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Recurrence of pelvic organ prolapse | 1 year
  Recurrence rate of cystocele, rectocele, uterine prolapse, or vaginal vault prolapse within 1 year after surgery

SECONDARY OUTCOMES:
The change of pad weight | 3 months
  The change of pad weight between baseline and 3 months after surgery for pelvic organ prolapse
The change of maximum urethral closure pressure | 3 months
  The difference of maximum urethral closure pressure between baseline and 3 months after surgery
Vaginal mesh erosion | 1 year
  Vaginal mesh erosion rate within 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, MD, PhD, Principal Investigator — Department of Obstetrics & Gynecology, National Taiwan University Hospital
Locations (1):
- Department of Obstetrics & Gynecology, National Taiwan University Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Derived] Chang TC, Hsiao SM, Chen CH, Wu WY, Lin HH. Clinical Outcomes and Urodynamic Effects of Tailored Transvaginal Mesh Surgery for Pelvic Organ Prolapse. Biomed Res Int. 2015;2015:191258. doi: 10.1155/2015/191258. Epub 2015 Nov 8. PMID 26634203